CLINICAL TRIAL: NCT05299723
Title: A Pilot Chronotherapeutic Intervention to Improve Sleep Following Acute Coronary Syndrome: The SleepWell Study
Brief Title: The SleepWell Study - Chronotherapeutic Intervention to Improve Sleep Following ACS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Ari Shechter, Assistant Professor of Medical Sciences, Columbia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AAAU0150; P30AG064198-02 (NIH)
Record Dates: First submitted 2022-03-15; First posted 2022-03-29 (Actual); Results first posted 2025-01-07 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2024-12

CONDITIONS: Sleep Disturbance; Insomnia; Acute Coronary Syndrome
Keywords: sleep; light therapy; chronotherapy; circadian; cardiovascular; insomnia; short sleep duration; intervention; acute coronary syndrome
MeSH Terms: conditions — Parasomnias; Sleep Initiation and Maintenance Disorders; Acute Coronary Syndrome

STUDY DESIGN:
Intervention Model Description: This will be a two-phase pilot study.
  Phase A of the study will be a single-arm open-label study of the home-based CC intervention in n=5 post-ACS patients. Please note that as Phase A is a single-arm open-label study, there will be no randomization of participants.
  Phase B of the study will be a parallel-arm randomized clinical trial (RCT) in which n=15 post-ACS patients will be randomized (using a 2:1 allocation) to active CC treatment or sleep hygiene education control group.
  The "Allocation" scheme below refers to Phase B.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Phase A - open label single-arm (Experimental): All Phase A participants randomized to the home-based CC intervention will be use a light visor to administer "bright light therapy" in the morning for 30 minutes after waking up (BLT), and use orange-colored glasses for "blue light blocking" at night from 8:00 pm until going to sleep (BLB).
  Interventions: Behavioral: BLT Intervention; Behavioral: BLB Intervention; Behavioral: Sleep Hygiene Education
- Phase B - active CC treatment (Experimental): For all Phase B participants randomized to the active CC group, BLT will occur each morning after awakening and will last for 30 minutes and BLB at night from 8:00 pm until going to sleep throughout the 4-week intervention period. Participants in the CC group will also receive a sleep hygiene education.
  Interventions: Behavioral: BLT Intervention; Behavioral: BLB Intervention; Behavioral: Sleep Hygiene Education
- Phase B - sleep hygiene education control group (Active Comparator): All Phase B participants randomized to the control group will receive a sleep hygiene education alone at the start of the 4 week monitoring period.
  Interventions: Behavioral: Sleep Hygiene Education

INTERVENTIONS:
Behavioral: BLT Intervention — BLT will be administered via a Luminette 3 light therapy visor. The Luminette 3 is a visor worn above the eyes containing light emitting diode (LEDs) emitting a blue-enriched white light reflecting to the retina at 1,000 lux via a holographic system in order to ensure correct penetration into the eye without impeding vision. This range of light and intensity is sufficient to synchronize the circadian clock.
  Other Names: Bright light therapy intervention
  Arms: Phase A - open label single-arm; Phase B - active CC treatment
Behavioral: BLB Intervention — BLB will be administered via orange lenses that filter out short-wavelength blue light, while allowing the other visible spectrum light to pass. The BLB lenses result in a reduction in melanopic irradiance (i.e., the light that affects sleep) of about 85%. The BLB lenses only make the overall light environment about 30% dimmer. Therefore, the BLB lenses are effective in blocking out most of the blue light in the visible environment that impacts sleep, but do not result in drastic overall dimming/darkening of the light environment.
  Other Names: Blue light blocking intervention
  Arms: Phase A - open label single-arm; Phase B - active CC treatment
Behavioral: Sleep Hygiene Education — The sleep hygiene education will consist of watching a sleep education video (background on the regulation of sleep, the impacts of insufficient sleep on mental and physical health, etc.) and a sleep hygiene video (providing overview of sleep hygiene approaches).

SUMMARY:
This two-phase pilot study will test the feasibility of a "combined chronotherapy" (CC) intervention consisting of morning bright light therapy (BLT) and evening blue light blocking (BLB), administered daily for 4 weeks in patients who experienced acute coronary syndrome (ACS). Phase A of the study will be a single-arm open-label study of the home-based CC intervention in 5 post-ACS patients. Phase B of the study will be a parallel-arm randomized clinical trial (RCT) in which 15 post-ACS patients will be randomized (using a 2:1 allocation) to active CC treatment or sleep hygiene education control group. In Phase A and Phase B, the primary aims are study feasibility, acceptability, appropriateness, and usability. In Phase B, the investigator will additionally assess whether the intervention engages its proposed proximal target mechanism - sleep.

DETAILED DESCRIPTION:
Survivors of acute medical events often experience psychological distress including post-traumatic stress disorder (PTSD). The goal of this project is to conduct preliminary testing of a chronotherapeutic intervention targeting disturbed sleep in survivors of ACS.

There are many ways to try and improve sleep. Some of these include taking medications or working with a trained sleep specialist. The goal of this research study is to investigate the usefulness of a new way of trying to improve sleep (an "intervention") that does not involve taking medications or working with a specialist or therapist. Chronotherapeutic interventions are non-pharmacologic approaches that target the circadian or sleep-wake cycle to improve behavioral or health outcomes. Light is the strongest external signal for the human circadian system and manipulations of the light environment (e.g., morning bright light exposure and evening light avoidance) are effective in improving sleep and mood.

Participants in Phase A of this study will be asked to use a light visor to administer light to the eye each morning (BLT component of the CC) and orange-colored glasses to block out short wavelength ("blue") light to the eye each night before going to bed (BLB component of the CC) for 4 weeks. Participants are also asked to wear an activity/sleep monitor throughout the 4-week period and complete questionnaires about their sleep. Participants will also receive a sleep hygiene education by watching educational videos.

In Phase B of the study, participants will be randomized to either the active CC intervention condition (consisting of both the BLT and BLB components along with sleep hygiene education) or a sleep hygiene education only control condition. Participants will be randomized in a 2:1 ratio to CC condition or control condition. All participants (i.e., those in the CC and control groups) will wear an activity/sleep monitor throughout the 4-week period and complete questionnaires about their sleep. There will also be a 3 month follow up after the end of the 4-week intervention period for both groups where we assess sleep outcomes.

ELIGIBILITY:
Patients will be eligible for PHASE A if they meet the following criteria

Inclusion Criteria:

1. 18 years of age or older,
2. can write, speak and read English,
3. provider and patient confirmed ACS,
4. ACS event occurred within the past 3 months, and
5. presence of insomnia symptoms based on the Insomnia Symptoms Questionnaire, or frequently (3-4 times per week) or always (5-7 times per week) experiencing short sleep duration of 6 hours or less per night.

Exclusion Criteria:

1. severe disabling chronic medical and/or psychiatric comorbidities determined on a case-by-case basis that prevent safe or adequate participation;
2. deemed unable to comply with the protocol (either self-selected or indicated during screening that s/he/they could not complete all requested tasks). This includes, but is not limited to, patients with a level of cognitive impairment indicative of dementia, patients with current alcohol or substance abuse, and patients with severe mental illness (e.g., schizophrenia);
3. unavailable for follow-up for reasons such as terminal illness and imminent plans to leave the United States (as we have migrant or mobile patients due to their citizenship and work issues);
4. Non-English speaking;
5. Lack of reliable phone or e-mail access;
6. History of bipolar disorder (manic episode can be triggered by BLT) or positive screen for bipolar disorder based on the Mood Disorder Questionnaire;
7. Eye disease including glaucoma or retinopathy (BLT contraindications);
8. Blindness;
9. Night shift work schedules;
10. taking any anti-depressant or anti-anxiety medications; and
11. taking other medications that increase sensitivity to light (by self-report).

Patients will be eligible for PHASE B if they meet the following criteria:

Inclusion Criteria:

1. 18 years of age or older,
2. can write, speak and read English or Spanish,
3. provider and patient confirmed ACS,
4. ACS event occurred within the past 3 months, and
5. presence of insomnia symptoms based on the Insomnia Symptoms Questionnaire, or frequently (3-4 times per week) or always (5-7 times per week) experiencing short sleep duration of 6 hours or less per night.

Exclusion Criteria:

1. severe disabling chronic medical and/or psychiatric comorbidities determined on a case-by-case basis that prevent safe or adequate participation;
2. deemed unable to comply with the protocol (either self-selected or indicated during screening that s/he/they could not complete all requested tasks). This includes, but is not limited to, patients with a level of cognitive impairment indicative of dementia, patients with current alcohol or substance abuse, and patients with severe mental illness (e.g., schizophrenia);
3. unavailable for follow-up for reasons such as terminal illness and imminent plans to leave the United States (as we have migrant or mobile patients due to their citizenship and work issues);
4. Non-English and non-Spanish speaking;
5. Lack of reliable phone or e-mail access;
6. History of bipolar disorder (manic episode can be triggered by BLT) or positive screen for bipolar disorder based on the Mood Disorder Questionnaire;
7. Eye disease including glaucoma or retinopathy (BLT contraindications);
8. Blindness;
9. Night shift work schedules;
10. taking any anti-depressant or anti-anxiety medications; and
11. taking other medications that increase sensitivity to light (by self-report).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2022-04-18 (Actual); Primary Completion 2024-02-27 (Actual); Study Completion 2024-06-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ari Shechter, PhD, Principal Investigator — Associate Professor of Medical Sciences
Locations (1):
- CUIMC, New York, New York, United States

REFERENCES:
- [Derived] Mendieta M, Cumella R, Fray N, Lopez-Veneros D, Hiti D, Franqui C, D'Agostino C, Kronish IM, Shechter A. Combined Chronotherapy for Poor Sleep Following Acute Coronary Syndrome: A Pilot Randomized Trial. J Circadian Rhythms. 2025 Feb 25;23:1. doi: 10.5334/jcr.250. eCollection 2025. PMID 40028185

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase A - Open Label Single-arm: All Phase A participants randomized to the CC used a light visor to administer "bright light therapy" in the morning for 30 minutes after waking up (BLT), and used orange-colored glasses for "blue light blocking" at night from 8:00 pm until going to sleep (BLB).
  BLT Intervention: BLT was administered via a Luminette 3 light therapy visor. The Luminette 3 is a visor worn above the eyes containing light emitting diode (LEDs) emitting a blue-enriched white light reflecting to the retina at 1,000 lux via a holographic system in order to ensure correct penetration into the eye without impeding vision. This range of light and intensity is sufficient to synchronize the circadian clock.
  BLB Intervention: BLB was administered via orange lenses that filter out short-wavelength blue light, while allowing the other visible spectrum light to pass. BLB lenses reduce melanopic irradiance (i.e., the light that affects sleep) of about 85%. BLB lenses only make the overall light environment about 30% dimmer. Therefore, the BLB lenses are effective in blocking out most of the blue light in the visible environment that impacts sleep, but do not result in drastic overall dimming/darkening of the light environment.
  Sleep Hygiene Education: The sleep hygiene education consisted of watching a sleep education video (background on the regulation of sleep, the impacts of insufficient sleep on mental and physical health, etc.) and a sleep hygiene video (overview of sleep hygiene approaches).
- Phase B - Active CC Treatment: For all Phase B participants randomized to the active CC group, BLT occurred each morning after awakening and lasted 30 minutes and BLB at night from 8:00 pm until going to sleep throughout the 4-week intervention period. Participants in the CC group also received sleep hygiene education.
  BLT Intervention: BLT was administered via a Luminette light therapy visor. Luminette is a visor worn above the eyes containing light emitting diode (LEDs) emitting a blue-enriched white light reflecting to the retina. This range of light and intensity is sufficient to synchronize the circadian clock.
  BLB Intervention: BLB was administered via orange lenses that filter out short-wavelength blue light, while allowing the other visible spectrum light to pass. The BLB lenses result in a reduction in melanopic irradiance (i.e., the light that affects sleep) of about 85%. The BLB lenses only make the overall light environment about 30% dimmer. Therefore, the BLB lenses are effective in blocking out most of the blue light in the visible environment that impacts sleep, but do not result in drastic overall dimming/darkening of the light environment.
  Sleep Hygiene Education: The sleep hygiene education consisted of watching a sleep education video (background on the regulation of sleep, the impacts of insufficient sleep on mental and physical health, etc.) and a sleep hygiene video (providing overview of sleep hygiene approaches).
Period: Overall Study
Arm/Group | Phase A - Open Label Single-arm | Phase B - Active CC Treatment | Phase B - Sleep Hygiene Education Control Group
Started | 4 | 10 | 5
Completed | 4 | 8 | 5
Not Completed | 0 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Population: Two patients from the Phase B CC intervention group withdrew from the study after randomization but before the start of study procedures.
Groups:
- Phase A - Open Label Single-arm: All Phase A participants randomized to the CC intervention used a light visor to administer "bright light therapy" in the morning for 30 minutes after waking up (BLT), and used orange-colored glasses for "blue light blocking" at night from 8:00 pm until going to sleep (BLB).
  BLT Intervention: BLT was administered via a Luminette light therapy visor. Luminette is a visor worn above the eyes containing light emitting diode (LEDs) emitting a blue-enriched white light reflecting to the retina. This range of light and intensity is sufficient to synchronize the circadian clock.
  BLB Intervention: BLB was administered via orange lenses that filter out short-wavelength blue light, while allowing the other visible spectrum light to pass. The BLB lenses result in a reduction in melanopic irradiance (i.e., the light that affects sleep) of about 85%. The BLB lenses only make the overall light environment about 30% dimmer. Therefore, the BLB lenses are effective in blocking out most of the blue light in the visible environment that impacts sleep, but do not result in drastic overall dimming/darkening of the light environment.
  Sleep Hygiene Education: The sleep hygiene education consisted of watching a sleep education video (background on the regulation of sleep, the impacts of insufficient sleep on mental and physical health, etc.) and a sleep hygiene video (providing overview of sleep hygiene approaches).
- Phase B - Active CC Treatment: For all Phase B participants randomized to the active CC group, BLT occured each morning after awakening and lasted for 30 minutes and BLB at night from 8:00 pm until going to sleep throughout the 4-week intervention period. Participants in the CC group also received a sleep hygiene education.
  BLT Intervention: BLT was administered via a Luminette light therapy visor. Luminette is a visor worn above the eyes containing light emitting diode (LEDs) emitting a blue-enriched white light reflecting to the retina. This range of light and intensity is sufficient to synchronize the circadian clock.
  BLB Intervention: BLB was administered via orange lenses that filter out short-wavelength blue light, while allowing the other visible spectrum light to pass. The BLB lenses result in a reduction in melanopic irradiance (i.e., the light that affects sleep) of about 85%. The BLB lenses only make the overall light environment about 30% dimmer. Therefore, the BLB lenses are effective in blocking out most of the blue light in the visible environment that impacts sleep, but do not result in drastic overall dimming/darkening of the light environment.
  Sleep Hygiene Education: The sleep hygiene education consisted of watching a sleep education video (background on the regulation of sleep, the impacts of insufficient sleep on mental and physical health, etc.) and a sleep hygiene video (providing overview of sleep hygiene approaches).
- Total: Total of all reporting groups
Arm/Group | Phase A - Open Label Single-arm | Phase B - Active CC Treatment | Phase B - Sleep Hygiene Education Control Group | Total
Number analyzed (Participants) | 4 | 10 | 5 | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.5 (6.8) | 60.9 (13.1) | 54.4 (17.3) | 59.7 (13.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 2 | 4
  Male | 4 | 8 | 3 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 3 | 2 | 8
  Not Hispanic or Latino | 0 | 6 | 3 | 9
  Unknown or Not Reported | 1 | 1 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 3 | 2 | 7
  White | 1 | 4 | 0 | 5
  More than one race | 0 | 1 | 1 | 2
  Unknown or Not Reported | 0 | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 4 | 10 | 5 | 19
Baseline Insomnia Severity Index score [Mean (Standard Deviation); unit: units on a scale] — The ISI consists of 5 questions rating presence and severity of insomnia using a 5-point Likert scale (0 through 4, with higher scores indicating worse severity). The ISI score is computed by adding up the score son each of the 5 questions. The score ranges from 0 to 28. Higher scores indicate worse severity insomnia symptoms
  units on a scale | 14 (6.2) | 11.4 (6.9) | 19.2 (3.4) | 13.5 (6.3)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Complete 100% of the Outcome Assessments at Study Conclusion
Description: The total number of participants who complete all endpoint questionnaire assessments will be documented and the proportion of participants who fully complete outcome assessments will be computed.
Time Frame: At end of 4-week intervention period
Measure: Count of Participants; unit: Participants
Arm/Group | Phase A - Open Label Single-arm | Phase B - Active CC Treatment | Phase B - Sleep Hygiene Education Control Group
Number analyzed (Participants) | 4 | 8 | 5
Participants | 4 | 7 | 5

2. Primary Outcome: Percentage of Participants Who Report Scores ≥4 for Their Final Rating of the Intervention's Feasibility
Description: Participants in Phase A and those participants in Phase B who were randomized to the intervention group will complete the Feasibility of Intervention Measure (FIM). The FIM is a 4-item questionnaire, with each question having a 5-point Likert scale (1=completely disagree to 5= completely agree). The score is calculated by adding up the selections on each of the 4 questions. The total score on the FIM can range from 4 to 20, with higher scores indicating greater feasibility of the intervention.
Time Frame: At end of 4-week intervention period
Population: Phase B participants in the sleep hygiene education group did not complete the FIM scale. Only those who used the intervention completed ratings.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase A - Open Label Single-arm | Phase B - Active CC Treatment | Phase B - Sleep Hygiene Education Control Group
Number analyzed (Participants) | 4 | 7 | 0
Participants | 4 | 5 | 0

3. Primary Outcome: Percentage of Participants Who Report Scores ≥4 for Their Final Rating of the Intervention's Acceptability
Description: Participants in Phase A and those participants in Phase B who were randomized to the intervention group will complete the Acceptability of Intervention Measure (AIM). The AIM is a 4-item questionnaire, with each question having a 5-point Likert scale (1=completely disagree to 5= completely agree). The score is calculated by adding up the selections on each of the 4 questions. The total score on the AIM can range from 4 to 20, with higher scores indicating greater acceptability of the intervention.
Time Frame: At end of 4-week intervention period
Population: Phase B participants in the sleep hygiene education group did not complete the AIM scale. Only those who used the intervention completed ratings.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase A - Open Label Single-arm | Phase B - Active CC Treatment | Phase B - Sleep Hygiene Education Control Group
Number analyzed (Participants) | 4 | 7 | 0
Participants | 2 | 4 | 0

4. Primary Outcome: Percentage of Participants Who Report Scores ≥4 for Their Final Rating of the Intervention's Appropriateness for Improving Sleep
Description: Participants in Phase A and those participants in Phase B who were randomized to the intervention group will complete the Intervention Appropriateness Measure (IAM). The IAM is a 4-item questionnaire, with each question having a 5-point Likert scale (1=completely disagree to 5= completely agree). The score is calculated by adding up the selections on each of the 4 questions. The total score on the IAM can range from 4 to 20, with higher scores indicating greater feasibility of the intervention.
Time Frame: At end of 4-week intervention period
Population: Phase B participants in the sleep hygiene education group did not complete the IAM scale. Only those who used the intervention completed ratings.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase A - Open Label Single-arm | Phase B - Active CC Treatment | Phase B - Sleep Hygiene Education Control Group
Number analyzed (Participants) | 4 | 7 | 0
Participants | 3 | 2 | 0

5. Primary Outcome: Percentage of Participants Who Report Total Scores ≥68 for Their Final Rating of the Intervention's Usability
Description: Participants in Phase A and those participants in Phase B who were randomized to the intervention group will complete the System Usability Scale (SUS). The SUS is a 10-item questionnaire with a 5-point Likert scale (1= strongly disagree to 5 = strongly agree). The score is calculated by subtracting 1 from each question's raw score then using the following equation: SUS = 2.5 (20 + [sum of scores on SUS1, SUS3, SUS5, SUS7, SUS9] - [sum of scores on SUS2, SUS4, SUS6, SUS8, SUS10]). The SUS total score can range from 0 to 100, with higher scores indicating better system usability of the intervention.
Time Frame: At end of 4-week intervention period
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Phase A - Open Label Single-arm | Phase B - Active CC Treatment | Phase B - Sleep Hygiene Education Control Group
Number analyzed (Participants) | 4 | 7 | 0
Participants | 4 | 7 | 0

6. Primary Outcome: Percentage of Who Report Administering the BLT Intervention on ≥50% of the Days Throughout the 4-wk Treatment Period
Description: Participants will complete a daily use log where the times of use of the intervention devices will be documented. Adherence to the protocol will be calculated as using the devices on ≥50% of days. The proportion of participants who meet adherence criteria at 4 week endpoint will be computed.
Time Frame: At end of 4-week intervention period
Population: Phase B participants in the sleep hygiene education group did not use the devices.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase A - Open Label Single-arm | Phase B - Active CC Treatment | Phase B - Sleep Hygiene Education Control Group
Number analyzed (Participants) | 4 | 8 | 0
Participants | 4 | 7 | 0

7. Secondary Outcome: Difference in the Total Score of Insomnia Severity Index
Description: This is to measure the baseline-to-study conclusion change in insomnia symptom severity. The range of values is 0-28, with higher values indicating worsened severity of insomnia symptoms. The total score is interpreted as follows: absence of insomnia (0-7); sub-threshold insomnia (8-14); moderate insomnia (15-21); and severe insomnia (22-28).
Time Frame: Baseline, 4 weeks
Measure: Mean (Standard Deviation); unit: pre-to-post change score on a scale
Arm/Group | Phase A - Open Label Single-arm | Phase B - Active CC Treatment | Phase B - Sleep Hygiene Education Control Group
Number analyzed (Participants) | 4 | 7 | 5
pre-to-post change score on a scale | -8.25 (7.3) | -5.7 (9.3) | -3.0 (4.6)

8. Secondary Outcome: Difference in the Total Global Score of Pittsburgh Sleep Quality Index
Description: This is to measure the baseline-to-study conclusion change in global sleep quality. The Pittsburgh Sleep Quality Index is a 19-item questionnaire that is completed by the participant. The score range is 0-21. Higher score indicates poorer sleep quality. A cutoff value of a total score > 5 is often used to indicate the presence of poor sleep quality.
Time Frame: Baseline, 4 weeks
Measure: Mean (Standard Deviation); unit: pre-to-post change score on a scale
Arm/Group | Phase A - Open Label Single-arm | Phase B - Active CC Treatment | Phase B - Sleep Hygiene Education Control Group
Number analyzed (Participants) | 4 | 7 | 5
pre-to-post change score on a scale | -5 (2.9) | -3.6 (3.8) | -3.2 (3.6)

9. Secondary Outcome: Difference in the Sleep Duration Item of the Pittsburgh Sleep Quality Index (i.e., Question #4).
Description: This is to measure the baseline-to-study conclusion change in self-reported sleep duration (hours spent asleep). Participants enter a value as a whole number in response to the question: "During the past month, how many hours of actual sleep did you get at night? (This may be different than the number of hours you spend in bed.)"
Time Frame: Baseline, 4 weeks
Measure: Mean (Standard Deviation); unit: pre-to-post change in hours
Arm/Group | Phase A - Open Label Single-arm | Phase B - Active CC Treatment | Phase B - Sleep Hygiene Education Control Group
Number analyzed (Participants) | 4 | 7 | 5
pre-to-post change in hours | 1 (1.1) | 1 (1.1) | 0.3 (1.6)

10. Primary Outcome: Percentage of Who Report Administering the BLT Intervention on ≥75% of the Days Throughout the 4-wk Treatment Period
Description: Participants will complete a daily use log where the times of use of the intervention devices will be documented. Adherence to the protocol will be calculated as using the devices on ≥75% of days. The proportion of participants who meet adherence criteria at 4 week endpoint will be computed.
Time Frame: At end of 4-week intervention period
Population: Phase B participants in the sleep hygiene education group did not use the devices.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase A - Open Label Single-arm | Phase B - Active CC Treatment | Phase B - Sleep Hygiene Education Control Group
Number analyzed (Participants) | 4 | 8 | 0
Participants | 4 | 5 | 0

11. Primary Outcome: Percentage of Who Report Administering the BLB Intervention on ≥50% of the Days Throughout the 4-wk Treatment Period
Description: as for outcome 6
Time Frame: At end of 4-week intervention period
Population: Phase B participants in the sleep hygiene education group did not use the devices.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase A - Open Label Single-arm | Phase B - Active CC Treatment | Phase B - Sleep Hygiene Education Control Group
Number analyzed (Participants) | 4 | 8 | 0
Participants | 4 | 8 | 0

12. Primary Outcome: Percentage of Who Report Administering the BLB Intervention on ≥75% of the Days Throughout the 4-wk Treatment Period
Description: as for outcome 10
Time Frame: At end of 4-week intervention period
Population: Phase B participants in the sleep hygiene education group did not use the devices.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase A - Open Label Single-arm | Phase B - Active CC Treatment | Phase B - Sleep Hygiene Education Control Group
Number analyzed (Participants) | 4 | 8 | 0
Participants | 4 | 7 | 0

ADVERSE EVENTS:
Time Frame: 4 weeks
Arm/Group | Phase A - Open Label Single-arm | Phase B - Active CC Treatment | Phase B - Sleep Hygiene Education Control Group
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/8 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/8 | 0/5
Other Adverse Events (participants affected / at risk) | 0/4 | 2/8 | 0/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase A - Open Label Single-arm (N=4) | Phase B - Active CC Treatment (N=8) | Phase B - Sleep Hygiene Education Control Group (N=5)
headache (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
eyestrain / eye sensitivity (Eye disorders) | 0 | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-07-28): https://cdn.clinicaltrials.gov/large-docs/23/NCT05299723/Prot_000.pdf
  • Statistical Analysis Plan (2023-07-28): https://cdn.clinicaltrials.gov/large-docs/23/NCT05299723/SAP_001.pdf